CLINICAL TRIAL: NCT01846832
Title: A Phase 3, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of TMC435 Plus Pegylated Interferon Alfa-2a and Ribavirin Administered for 12 Weeks in Treatment-Naïve Subjects With Chronic Genotype 1 or Genotype 4 HCV Infection
Brief Title: A Study of TMC435 Plus Pegylated Interferon Alfa-2a and Ribavirin in Participants With Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100981; TMC435HPC3014 (Other: Janssen-Cilag International NV); 2012-004905-29 (EudraCT Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C, Chronic; Infection
Keywords: Hepatitis C, Chronic; Infection; Triple therapy; TMC435; simeprevir; Pegylated interferon alfa-2a (PegIFNα-2a); ribavirin (RBV); PEGASYS; COPEGUS
MeSH Terms: conditions — Hepatitis C, Chronic; Infections | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMC435 + PegIFNα-2a + RBV (Experimental): TMC435 will be administered as triple therapy with pegylated interferon alfa-2a (PegIFNα-2a) and ribavirin (RBV).
  Interventions: Drug: TMC435; Drug: Pegylated interferon alfa-2a (PegIFNα-2a); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: TMC435 — 150 mg taken orally (by mouth) as a capsule with food once daily for 12 weeks.
Drug: Pegylated interferon alfa-2a (PegIFNα-2a) — 180 mcg administered according to the manufacturer's prescribing information as a 0.5 mL subcutaneous (under the skin) (SC) injection once a week in the morning or evening for up to 24 weeks.
  Other Names: Pegasys
Drug: Ribavirin (RBV) — 1000 mg or 1200 mg administered according to the manufacturer's prescribing information for up to 24 weeks. If the participant's baseline body weight is < 75 kg, the total daily dose of RBV will be 1000 mg, administered orally (by mouth) as 400 mg (2 tablets of 200 mg, intake with food) in the morning and 600 mg (3 tablets of 200 mg, intake with food) in the evening. If the baseline body weight is > or = 75 kg, the total daily dose will be 1200 mg, administered as 600 mg in the morning and evening (3 tablets of 200 mg per intake, with food).
  Other Names: Copegus

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability, and safety of 12-weeks of treatment with TMC435 plus pegylated interferon alfa-2a (PegIFNα-2a) and ribavirin (RBV) in previously untreated adult participants with genotype 1 or genotype 4 chronic Hepatitis C Virus (HCV) infection.

DETAILED DESCRIPTION:
This is a multicenter, international study where all participants will receive triple therapy with the following 3 medications: TMC435 also referred to as simeprevir (formerly known as TMC435350) which is an investigational medication in development for the treatment of chronic hepatitis C virus (HCV) infection, pegylated interferon alfa-2a (PegIFNα-2a), and ribavirin (RBV). PegIFNα-2a and RBV are commercially available therapies for HCV infection. Participants will receive treatment with TMC435, PegIFNα-2a, and RBV for 12 weeks. If blood levels of HCV ribonucleic acid (RNA) monitored at Weeks 2, 4, and 8 are below 25 IU/mL, all treatment will be stopped at Week 12. If HCV RNA values are above 25 IU/mL at Weeks 2, 4, or 8, treatment with PegIFNα-2a and RBV will continue for an additional 12 weeks (up to Week 24) unless protocol-specified stopping criteria are met at Week 4 or 12, at which time all treatment will be discontinued. The study will be conducted in 3 phases: a screening phase of maximum 6 weeks, a treatment phase extending from Day 1 (baseline) up to 12 or 24 weeks depending on the response to treatment, and a posttreatment follow-up period of 24 weeks after the participant's last planned dose of study drug. The duration of the participation (excluding screening phase) for each participant will vary between 36 and 48 weeks, depending on the response to treatment. Blood samples for laboratory analysis will be obtained from participants at protocol-specified time points during the study and participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* treatment-naïve with confirmed chronic Hepatitis C Virus (HCV) infection
* liver biopsy performed within 2 years prior to screening or non-invasive confirmation of the liver disease stage (by transient elastography) performed within 6 months prior to screening
* liver disease stage equivalent to Metavir Score F0-F2 (no fibrosis, or portal fibrosis without or with few septa)

Exclusion Criteria:

-Participants with advanced liver disease equivalent to Metavir score F3-F4 (bridging fibrosis or cirrhosis), with hepatic decompensation, with any liver disease of non-HCV etiology, and/or with a non-genotype 1 or non-genotype 4 hepatitis C, hepatitis B or HIV co-infection will be excluded from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The proportion (percentage) of participants infected wtih genotype 1 HCV with a sustained virologic response 12 weeks after planned end of treatment (SVR12) | Week 24
  Participants are considered to have reached SVR12 if at the actual end of treatment hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 25 IU/mL undetectable, AND at the time point of SVR12 (i.e., 12 weeks after the planned end of treatment [EOT]), HCV RNA levels < 25 IU/mL undetectable.

SECONDARY OUTCOMES:
The proportion (percentage) of participants infected wtih genotype 4 HCV with a sustained virologic response 12 weeks after planned end of treatment (SVR12) | Week 24
  See SVR12 defined above.
The proportion (percentage) of participants who achieve rapid virologic response (RVR) | Week 4
  Rapid virologic response (RVR) defined as hepatitis C virus (HCV) ribonucleic acid (RNA) < 25 IU/mL undetectable measured 4 weeks after start of treatment. RVR will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants who achieve virologic response at Week 2 (W2VR) | Week 2
  Virologic response at Week 2 (W2VR) defined as hepatitis C virus (HCV) ribonucleic acid (RNA) < 25 IU/mL (detectable or undetectable) measured 2 weeks after start of treatment. W2VR will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with sustained virologic response 24 weeks after planned end of treatment (SVR24) | Week 48
  Participants are considered to have reached SVR24 if at the actual end of treatment hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 25 IU/mL undetectable, AND at the time point of SVR24 (i.e., 24 weeks after the planned end of treatment [EOT]) HCV RNA levels < 25 IU/mL undetectable. SVR24 will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with sustained virologic response 12 weeks after planned end of treatment (SVR12) | Week 24
  SVR12 (defined above) will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with > or = 2 log decrease in hepatitis C virus (HCV) RNA at each time point | Up to Week 48
  To be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with hepatitis C virus (HCV) RNA < 25 IU/mL undetectable at each time point | Up to Week 48
  To be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with viral breakthrough | Up to Week 48
  Viral breakthrough is a confirmed increase of > 1 log10 IU/mL in hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached, or a confirmed HCV RNA level of > 100 IU/mL in participants whose HCV RNA levels had previously been below the limit of quantification (< 25 IU/mL detectable) or undetectable (< 25 IU/mL undetectable) while on study treatment. Viral breakthrough will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
The proportion (percentage) of participants with viral relapse | Up to Week 48
  Participants are considered to have a viral relapse if at actual end of treatment hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 25 IU/mL undetectable, AND during the follow-up period HCV RNA levels > or = 25 IU/mL. Viral relapse will be assessed for all participants per assigned total treatment duration and per HCV genotype (separately).
Change from Baseline in the Hepatitis C Treatment Symptom & Impact Questionnaire (HCV SIQ) symptom and impact scores | Day 1 and at each study visit up to Week 48
  The HCV SIQ asks participants to rate 26 symptoms associated with HCV or its treatment and how symptoms impacted the participants' life during the prior week. This questionnaire provides a simple tool for monitoring symptoms during HCV treatment and follow-up. To be assessed in participants with genotype 1 or genotype 4 HCV infection for both genotypes combined (subanalyses for each genotype separately will also be done).
Change from Baseline in The Fatigue Severity Scale (FSS) total score | Day 1 and at each study visit up to Week 48
  The FSS will be used to document fatigue severity and impact of fatigue on participants' daily lives. To be assessed in participants with genotype 1 or genotype 4 HCV infection for both genotypes combined (subanalyses for each genotype separately will also be done).
Change from Baseline in The Center for Epidemiologic Studies Depression Scale (CES-D) score | Day 1 and at each study visit up to Week 48
  The CES-D is a brief assessment that asks participants to rate how often in the past week they experienced 20 symptoms associated with depressive illness, will be used to assess depressive symptom severity. To be assessed in participants with genotype 1 or genotype 4 HCV infection for both genotypes combined (subanalyses for each genotype separately will also be done).
Change from Baseline in The Work Productivity and Activity Index (WPAI) for Hepatitis C missed work time, daily activity impairment, and productivity scores | Day 1 and at each study visit up to Week 48
  The (WPAI) will be used to measure the impact of HCV on time missed from work (absenteeism), reduced performance while at work (productivity impairment), and impairment in daily activities without regard to employment status. To be assessed in participants with genotype 1 or genotype 4 HCV infection for both genotypes combined (subanalyses for each genotype separately will also be done).
Change from Baseline in The EuroQol 5 Dimension (EQ5D) Visual Analog Scale (VAS) valuation index, and Descriptive System scores | Day 1 and at each study visit up to Week 48
  The EQ-5D questionnaire is an instrument designed to assess overall health status using 5 health dimension scores (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a "thermometer" visual analog scale (VAS) ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). To be assessed in participants with genotype 1 or genotype 4 HCV infection for both genotypes combined (subanalyses for each genotype separately will also be done).
The proportion (percentage) of participants with normalized alanine aminotransferase (ALT) levels | Up to Week 48
  To be assessed in participants with genotype 1 or genotype 4 HCV infection (separately by genotype)
Change from Screening in liver disease stage assessment | Week -6; Week 48
  To be assessed in participants with genotype 1 or genotype 4 HCV infection (separately by genotype).
The number of participants reporting adverse events as a measure of safety and tolerability | Up to Week 48
  All participants will be monitored throughout the study for the occurrence of adverse events including psychiatric symptoms, anemia, hyperglycemia (elevated glucose levels), disturbances in serum creatinine levels (a measure of renal [kidney] safety), decreased White Blood Cell (WBC) Count, decreased Platelet Count (ability of the blood to clot), and thyroid abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: JJanssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (20):
- Austria (2):
  - Linz
  - Vienna
- Belgium (2):
  - Brussels
  - Edegem
- France (4):
  - Clichy
  - Limoges
  - Orléans
  - Saint-Laurent-du-Var
- Germany (5):
  - Berlin
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Würzburg
- Riyadh, Saudi Arabia
- Spain (4):
  - Barcelona
  - Madrid
  - Valencia
  - Valme
- United Kingdom (2):
  - Glasgow
  - London

REFERENCES:
- [Derived] Asselah T, Moreno C, Sarrazin C, Gschwantler M, Foster GR, Craxi A, Buggisch P, Sanai F, Bicer C, Lenz O, Van Dooren G, Nalpas C, Lonjon-Domanec I, Schlag M, Buti M. Efficacy of a 12-Week Simeprevir Plus Peginterferon/Ribavirin (PR) Regimen in Treatment-Naive Patients with Hepatitis C Virus (HCV) Genotype 4 (GT4) Infection and Mild-To-Moderate Fibrosis Displaying Early On-Treatment Virologic Response. PLoS One. 2017 Jan 5;12(1):e0168713. doi: 10.1371/journal.pone.0168713. eCollection 2017. PMID 28056030
- [Derived] Asselah T, Moreno C, Sarrazin C, Gschwantler M, Foster GR, Craxi A, Buggisch P, Ryan R, Lenz O, Scott J, Van Dooren G, Lonjon-Domanec I, Schlag M, Buti M. An Open-Label Trial of 12-Week Simeprevir plus Peginterferon/Ribavirin (PR) in Treatment-Naive Patients with Hepatitis C Virus (HCV) Genotype 1 (GT1). PLoS One. 2016 Jul 18;11(7):e0158526. doi: 10.1371/journal.pone.0158526. eCollection 2016. PMID 27428331
- See also: A Phase 3, Open-Label Study to Evaluate the Safety and Efficacy of TMC435 plus Pegylated Interferon alfa-2a and Ribavirin Administered for 12 Weeks in Treatment-Naïve Subjects with Chronic Genotype 1 or Genotype 4 HCV Infection — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3649&filename=(CR100981)_CSR%20.pdf